CLINICAL TRIAL: NCT06453720
Title: Optimizing Patient Treatment Involving Microbiome Integration for Specialized Therapeutics
Brief Title: Predicting IBD Treatment Outcomes With Gut Microbiome Analysis
Acronym: OPTIMIST
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: IBD Centre of BC (Unknown); GI Research Institute (Unknown); Pacific Gastroenterology Associates (Unknown)
Responsible Party: Principal Investigator, Genelle Lunken, Assistant Professor, University of British Columbia
Other Study IDs: H23-02927
Record Dates: First submitted 2024-05-22; First posted 2024-06-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
Keywords: IBD; Crohn Disease; Biologic Therapy; Immunology; Gastrointestinal Tract
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mucosal washings, intestinal biopsies, whole blood, serum, plasma, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Crohn's disease: The study will include 75 consenting patients with Crohn's disease, varying in levels of severity depending on assigned SES-CD scoring from their gastroenterologist. These patients will be undergoing routine colonoscopy as per their normal care routine, with this study not requiring additional scheduling commitments. Blood, mucosal washing, and intestinal biopsy samples will be collected during routine colonoscopy procedure. The patient will have the option to collect a stool sample the day before their colonoscopy and bring it to their appointment. They will also receive a sample collection kit during their appointment to collect their next required stool sample in two weeks after their scope.
  Interventions: Procedure: Colonoscopy
- Patients without inflammatory bowel disease: The study will include 25 non-IBD age and sex-matched controls to compare data alongside the CD patients. These patients will be undergoing routine colonoscopy as per their normal colon screening routine, with this study not requiring additional scheduling commitments. Blood, mucosal washing, and intestinal biopsy samples will be collected during routine colonoscopy procedure. The patient will have the option to collect a stool sample the day before their colonoscopy and bring it to their appointment. They will also receive a sample collection kit during their appointment to collect their next required stool sample in two weeks after their scope.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — A colonoscopy will be performed as part of routine clinical care for all participants, with the study not requiring any additional scheduling commitments outside of routine care.

SUMMARY:
The goal of this prospective observational study is to determine if specific microbiome signatures can predict therapeutic responses in adult patients with Crohn's disease (CD), a form of inflammatory bowel disease (IBD), living in British Columbia, Canada. The main questions this study seeks to answer are:

1. Can microbiome signatures across different sample types (fecal, intestinal washings, and intestinal epithelial biopsies) predict response to therapy in CD?
2. How do microbiome profiles differ between active and quiescent CD and non-IBD controls?

Researchers will compare microbiome signatures in patients with active and inactive CD as well as non-IBD controls to see if there are any microbial signatures that predict response to therapy.

Participants will:

1. Provide fecal and blood samples.
2. Undergo intestinal washings and intestinal epithelial biopsy specimens taken during routine colonoscopy.
3. Participate in a longitudinal follow-up over 12 months to monitor clinical, biochemical, and endoscopic responses to therapy.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic and relapsing inflammatory condition affecting the gastrointestinal (GI) tract. The study aims to evaluate microbiome profiles (bacteriome, and mycobiome) across three different sample types (fecal, intestinal washings, and intestinal epithelial biopsies) in a cohort of adult patients with Crohn's disease (CD) living in British Columbia, Canada, and investigate whether a microbial signature may predict response to IBD therapy.

Aims:

1. Determine microbiome signatures, across different sample types, in quiescent and active disease for patients with CD living in BC, Canada.
2. Evaluate whether fecal, mucosal, and/or intestinal epithelial biopsy microbiome signatures can predict response to therapy.

Methods

Study Design:

Phase 1: A cross-sectional pilot study to evaluate the microbiome in patients with IBD (with active and quiescent disease) and in non-IBD controls.

Primary Outcome: Compare results of microbial analyses (including bacteriome and mycobiome) across three different sample types: intestinal washings and intestinal epithelial biopsy specimens taken during colonoscopy, as well as fecal samples.

Secondary Outcomes: Investigate correlations between the microbial analyses across different sample types and disease activity in CD. Compare the difference in microbial analyses within each sample type between active and quiescent CD as well as non-IBD patients. Investigate if fecal microbiome composition and function 2 weeks after bowel preparation is comparable to pre-bowel preparation fecal microbiome in a subset of patients with CD.

Phase 2: A longitudinal observational study with a 12-month follow-up.

Primary Outcome: Identify if there are any microbial signatures that predict response to therapy in patients with active disease requiring escalated therapy, assessed clinically and biochemically after induction (12-16 weeks) and at 12 months (+/- 3 months).

Secondary Outcomes: Compare the sensitivity and specificity of microbial analyses from each sample type in predicting response to therapy.

ELIGIBILITY:
Inclusion Criteria:

CD patients:

* Adult patients ≥19 years old and ≤ 80 years old.
* CD with distal small bowel and/or colonic involvement that is endoscopically assessable with colonoscopy.
* Undergoing colonoscopy as part of routine clinical care.
* Active or quiescent disease.
* Active disease will be defined as a simple endoscopic score for CD (SES-CD).
* Quiescent disease is defined as an SES-CD <3.
* Mild active disease will be defined as a SES-CD of 3-6, or 3 with isolated ileal CD.
* Moderate/severe active disease will be defined as a simple endoscopic score for CD (SES-CD) ≥ 7 or ≥ 4 for isolated ileal CD.

Non-IBD controls:

* Adult patients ≥ 19 years old and ≤ 80 years old.
* Undergoing colonoscopy as part of colorectal screening.

Exclusion Criteria:

CD patients:

* Active perianal CD - defined as collection on MRI or clinically active fistula (i.e., draining fistula).
* Proximal small bowel (defined as not endoscopically assessable by colonoscopy) or isolated upper GI CD.
* Colectomy or Proctocolectomy.
* Pouch, J-Pouch or Reversed pouch surgery.
* Short Bowel Syndrome (SBS) diagnosis.
* Antibiotics in the last 2 months for any indication.
* Gastroenteritis or travel outside of Canada and the United States in the last month.
* Colorectal cancer, high-grade dysplasia or a polyp ≥2cm diagnosed at baseline endoscopy.
* Pregnant or breastfeeding.
* Bowel resection within the preceding 4 months.
* Primary sclerosing cholangitis.

Non-IBD controls:

* Found to have inflammation (deemed by endoscopist) at colonoscopy.
* History of IBD in 1st degree relative.
* Antibiotics in the last 2 months.
* Gastroenteritis or travel outside of Canada and the United States in the last month.
* Pregnant or breastfeeding.
* Previous bowel surgeries.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to have 75 CD patients complete phase 1 and 2, and 25 non-IBD controls to complete phase 1 only.
  Patient grouping for recruitment is as follows:
  * Group 1: 25 CD in endoscopic remission (SES-CD score <3).
  * Group 2: 25 CD with moderate to severe endoscopically active disease (SES-CD ≥ 7 or ≥ 4 for isolated ileal CD).
  * Group 3: 25 CD with mildly endoscopically active disease (SES-CD of 3-6, or 3 with isolated ileal CD).
  * Group 4: 25 age, sex-matched non-IBD controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Compare results of microbial analyses (including bacteriome and mycobiome) across three different sample types: intestinal washings and intestinal epithelial biopsy specimens taken during colonoscopy as well as fecal samples. | 24 months
  Microbial analyses that will be undertaken for each sample type are as follows:
  Stool:
  * Metagenomics (Shotgun sequencing, ITS sequencing for fungal analysis)
  * Metaproteomics and metabolomics (Host, microbial, and dietary protein analysis, microbial metabolite analysis)
  * Anaerobic culturing (Simulate gut environment, use dietary substrates to target key microbes)
  Biopsy specimens:
  * Organoid culturing (In vitro gut model analysis, epithelial-microbiome analysis, mucin production analysis)
  * RNA-seq, transcriptomics (Gene expression profiling analysis, disease marker identification)
  * Metagenomics
  * Metaproteomics and metabolomics
  Intestinal washings:
  * Mucin analysis (Glycoprotein analysis)
  * Metagenomics
  * Metaproteomics and metabolomics
In patients with active Crohn's disease, where a decision is made to escalate therapy after the index endoscopy, identify if there are any microbial signatures that predict response to therapy after induction (12 - 16 weeks). | 24 months
  * Clinical Response: Defined based on changes in clinical symptoms as per standardized clinical scoring systems (SES-CD).
  * Biochemical Response: Assessed through C-reactive protein (CRP) levels and fecal calprotectin, two biomarkers that indicate inflammation or disease activity.
  The Simple Endoscopy Score for Crohn's Disease (SES-CD) is an objective clinical assessment of the severity of a patient's Crohn's disease. A higher score means more severe disease activity. The three severity classes of SES-CD scoring are as follows:
  * Endoscopic remission (SES-CD <3).
  * Moderate to severe endoscopically active disease (SES-CD ≥ 7 or ≥ 4 for isolated ileal CD).
  * Mild endoscopically active disease (SES-CD of 3-6, or 3 with isolated ileal CD).
In patients with active Crohn's disease, where a decision is made to escalate therapy after the index endoscopy, identify if there are any microbial signatures that predict sustained response to therapy at 12 Months (+/- 3 months). | 24 months
  * Clinical Response: Continuation or improvement in clinical symptoms as measured by standardized clinical scoring systems (SES-CD).
  * Biochemical Response: Persistent normalization or improvement in CRP levels and fecal calprotectin.
  * Endoscopic Response: Improvement or healing of mucosal lesions as observed during endoscopic examination, assessed by validated clinical scoring systems (SES-CD).

SECONDARY OUTCOMES:
Investigate the correlations between the microbial analyses across different sample types and disease activity in CD. | 24 months
  Correlation Analysis: Statistical measures will be used to assess the strength and direction of the relationship between microbial composition in different sample types (intestine washings, intestinal biopsy, fecal samples) and disease activity in CD.
  Disease Activity Measures: Disease activity will be assessed using the modified Harvey-Bradshaw Index, biochemical markers (CRP, fecal calprotectin), and endoscopic findings (SES-CD).
Compare the difference in microbial analyses within each sample type between active and quiescent CD as well as non-IBD patients. | 24 months
  Assessments:
  1. Microbial Diversity Metrics:
  * Alpha-diversity Metrics:
    * Shannon index
    * Inverse Simpson diversity index
    * Chao1
  * These metrics will be used to compare microbial diversity within each sample type between active and quiescent CD patients, as well as non-IBD patients.
Compare the difference in microbial analyses within each sample type between active and quiescent CD as well as non-IBD patients. | 24 months
  Assessments:
  Differential Abundance Analysis: Differential abundance analysis will be performed using generalized linear models to identify specific microbial taxa that are significantly different between active and quiescent CD patients, and non-IBD patients within each sample type.
Investigate, in a subset of patients with CD, if fecal microbiome composition and function 2 weeks after bowel preparation is comparable to pre-bowel preparation fecal microbiome. | 24 months
  Assessments:
  Comparison of Microbial Composition: Beta-diversity metrics (Bray-Curtis dissimilarity, Jaccard index) and phylogenetic-dependent distance metrics (weighted and unweighted UniFrac) will be calculated, and subsequent clustering will be applied using a principal coordinate analysis (PCoA). To test for overall microbiome differences, a PERMANOVA test will be applied. The Benjamini-Hochberg method will be applied to control for the false discovery rate.
Investigate, in a subset of patients with CD, if fecal microbiome composition and function 2 weeks after bowel preparation is comparable to pre-bowel preparation fecal microbiome. | 24 months
  Assessments:
  Functional Analysis: Functional profiling of the microbiome will be conducted to assess if there are any changes in the metabolic pathways and functions of the microbiome between pre- and post-bowel preparation samples in the subset of CD patients.
Compare the sensitivity of the microbial analyses from each sample type in their prediction of response to therapy. | 24 months
  Sensitivity of Microbial Analyses:
  * Using predictive models developed from microbial and statistical analyses, the sensitivity of microbial analyses from each sample type will be evaluated.
  * Sensitivity will be reported as the proportion of true positives correctly identified by the analysis.
Compare the specificity of the microbial analyses from each sample type in their prediction of response to therapy. | 24 months
  Specificity of Microbial Analyses:
  * Predictive models will also be used to evaluate the specificity of microbial analyses from each sample type.
  * Specificity will be reported as the proportion of true negatives correctly identified by the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- GI Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Massaro CA, Meade S, Lemarie FL, Kaur G, Bressler B, Rosenfeld G, Leung Y, Williams AJ, Lunken G. Gut microbiome predictors of advanced therapy response in Crohn's disease: protocol for the OPTIMIST prospective, longitudinal, observational pilot study in Canada. BMJ Open. 2025 Mar 13;15(3):e094280. doi: 10.1136/bmjopen-2024-094280. PMID 40082000